CLINICAL TRIAL: NCT04883684
Title: A Multi-institutional Study to Evaluate Patient Satisfaction of the Personal Health Record Management Platform for Chronic Patients in Emergency Department Based on Actual Demand
Brief Title: A Study to Evaluate Satisfaction of the Personal Health Record Platform for Chronic Patients in Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Taerim Kim, Clinical Assistant Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-03-019-006
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Emergencies, Chronic Disease
MeSH Terms: conditions — Emergencies; Chronic Disease | interventions — Emergency Service, Hospital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients(Care givers) (Experimental): 1. 400 patients(caregivers) are enrolled and use the personal health wallet service (Personal Health Records service).
  2. They fill out questionnaire to evaluate the service
  3. Some of them are invited for an in-depth interview.
  Interventions: Other: Personal health wallet service for Chronic Patients in Emergency Department

INTERVENTIONS:
Other: Personal health wallet service for Chronic Patients in Emergency Department — Patients(caregivers) will be provided the personal health wallet service and evaluate the effectiveness and satisfaction for the service.

SUMMARY:
The investigators developed the service showing patient health record altogether which is managed by each hospital separately and recording the patient health information based on mobile application. This study is a multi-centered study involving two hospitals, providing services to patients, care givers and medical staffs. After the participants use this service, the investigators evaluate the effectiveness and satisfaction of this service through questionnaires and in-depth interviews.

DETAILED DESCRIPTION:
<Background> Emergency situations for chronic patients are increasing due to aging, eating habits and lifestyle changes. For chronic patients, comprehensive health records and utilization are important for health care and emergency situations. In particular, in the event of an emergency, information on the patient's personal health records, such as recent surgery records, disease history, prescription and dosage history is needed immediately, but it is difficult to check separately for each hospital. In addition, in emergencies, it may take more time for proper treatment to take place if patients themselves cannot directly talk about their medication or past surgical history, or if they are unable to communicate with patients. Recently, conditions have been prepared for the collection and utilization of personal health record information due to changes in policy and technology environment, making it possible to provide services for emergency patients with chronic diseases.

<Objective> To establish a service for collection and utilization of medical records (care, examination, surgery, prescription records) and PGHD for chronic patients and to evaluate its effectiveness.

<Design> Mixed methods study (questionnaires and interview)

<Setting> At the Samsung Medical Center and the Dong-A Medical Center.

<Enrollment> 400 patients(care givers)

<Intervention>

1. 400 patients(care givers) are enrolled and use the personal health wallet service. (Personal Health Record service)
2. The participants fill out questionnaire to evaluate the service
3. Some of them are invited for an in-depth interview.

ELIGIBILITY:
<Inclusion Criteria>

* A chronic patient (or his or her care giver) who visits the emergency department and has a plan to visit outpatient or other hospitals in one month of the visiting emergency department.
* Adults over 19 years old.
* Those who voluntarily agreed to participate in the research

<Exclusion Criteria>

* Anyone who disagrees with this study
* Patients who are not conscious when leaving the emergency room, patients who are not aware of or are not aware of their orientation, patients who are not aware of their level of awareness, or people who are in shock or in deep shutdown situations) (Even in the above cases, caregivers can be included in the clinical trial target if they are present. )

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
SUS(System Usability Scale)-based assessment of patients or care givers satisfaction using personal health wallet service. | The day of the enrollment of the study
  SUS(System Usability Scale)-based assessment of patients or care givers satisfaction using personal health wallet service. SUS consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. Its score range is 0~100 and the higher the score, the higher the satisfaction level.
SUS(System Usability Scale)-based assessment of patients or care givers satisfaction using personal health wallet service. | 2 weeks after the enrollment
  SUS(System Usability Scale)-based assessment of patients or care givers satisfaction using personal health wallet service. SUS consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. Its score range is 0~100 and the higher the score, the higher the satisfaction level.
SUS(System Usability Scale)-based assessment of patients or care givers satisfaction using personal health wallet service. | 4 weeks after the enrollment
  SUS(System Usability Scale)-based assessment of patients or care givers satisfaction using personal health wallet service. SUS consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. Its score range is 0~100 and the higher the score, the higher the satisfaction level.
SUS(System Usability Scale)-based assessment of patients or care givers satisfaction using personal health wallet service. | 8 weeks after the enrollment
  SUS(System Usability Scale)-based assessment of patients or care givers satisfaction using personal health wallet service. SUS consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. Its score range is 0~100 and the higher the score, the higher the satisfaction level.

SECONDARY OUTCOMES:
A qualitative study on the satisfaction of patients or care givers through interviews | through study completion, an average of 3 months"
  A qualitative study on the satisfaction of patients or caregivers through interviews
A quantitative or qualitative study on the log data of the application | through study completion, an average of 3 months"
  A quantitative or qualitative study on the log data of the application

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea